CLINICAL TRIAL: NCT01806792
Title: For 4 Months, the Multi Center, Double Blinded, Randomized, Active Controlled, Comparative Clinical Study to Assess the Efficacy and the Safety to Improvement Effect of Vit.D of Risenex Plus M Tablet in Patients With In Post-menopausal Women Osteoporosis
Brief Title: Post-menopausal Women Osteoporosis(Phase III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_RSNPM_301
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Postmenopausal Women Osteoporosis
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risendronate and Cholecalciferol combination (Experimental): risedronate 150mg and cholecalciferol 30,000 IU 1 tablet + Placebo(for risedronate 150mg) 1 tablet by once a month.
  Interventions: Drug: risedronate combine; Drug: Placebo(for Risedronate)
- Risedronate (Active Comparator): risedronate 150mg 1 tablet + Placebo(for risedronate 150mg and cholecalciferol 30,000 IU) 1 tablet by once a month.
  Interventions: Drug: Risedronate; Drug: Placebo(for risedronate combine)

INTERVENTIONS:
Drug: risedronate combine
  Other Names: - Other name : Risenex M(risedronate 150mg and cholecalciferol 30,000 IU combined)
  Arms: Risendronate and Cholecalciferol combination
Drug: Risedronate
  Other Names: Other name : Actonel(Risedronate 150mg)
  Arms: Risedronate
Drug: Placebo(for Risedronate)
  Other Names: once a month
  Arms: Risendronate and Cholecalciferol combination
Drug: Placebo(for risedronate combine)
  Other Names: once a month
  Arms: Risedronate

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of Risedronate, cholecalciferol combination tablet in patients with Osteoporosis

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and the safety of Monthly Risedronate with cholecalciferol on 25 Hydroxyvitamin D level and bone markers patients with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. women osteoporosis
2. patients with a diagnosis of Postmenopausal over 6 Months if they had a bone mineral density T-score of < -2.5 at the mean lumbar spine (L1-4), femoral neck, or total, or a T-score of < -1.0 with radiologic evidence of at least one vertebral fracture. Menopause was defined as no natural menses for at least 1 year and a serum FSH level > 40 IU/L, with a reported hysterectomy
3. low levels of 25(OH)D > 9 ng/mL
4. patients who give written consent of agreement to voluntarily participate in the clinical study
5. patients who can read and understand written instructions

Exclusion Criteria:

1. patients who had contraindications to oral bisphosphonates, such as esophageal strictures
2. ALT, AST ≥ 2×UNL and Serum Creatinine ≥ 1.5×UNL
3. low levels of 25(OH)D (less than 9 ng/mL).
4. Previous use of oral bisphosphonates and vitamin D were allowed, but a washout period was needed, depending on the duration of treatment. Two-year washout periods were needed for bisphosphonate users and 3-6-month periods were required for vitamin D users of > 200 IU.
5. drug administration after diagnosing as alcoholic or psychical disease
6. patients whom the investigators judge as improper to participate in this clinical trial 7)13.patients who have experience to participate in other clinical trial within 30 days prior to study participation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
proportion of patients with 25(OH)D level < 20 ng/mL at 16 weeks. | 16 weeks form first drug adminstration.

SECONDARY OUTCOMES:
proportion of patients with 25(OH)D level < 9 ng/mL at 16 weeks, change of 25(OH)D level and Bone Markers. | 16 weeks form first drug administration.
  Secondary end point is :
  1. proportion of patients with 25(OH)D level < 9 ng/mL at 16 weeks
  2. change of 25(OH)D level
  3. change of BSAP
  4. change of CTX
  5. change of Ca
  6. change of phosphorous
  7. change of PTH
  8. change of 8-foot walking test, Sit-To-Stand test

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Moo Park, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-ang university hospital, Seoul, South Korea